CLINICAL TRIAL: NCT01537861
Title: A Pilot Study of G-CSF to Disrupt the Bone Marrow Microenvironment in Bortezomib-, Carfilzomib-, or IMID-Refractory Multiple Myeloma
Brief Title: Filgrastim in Treating Patients With Bortezomib-, Carfilzomib-, or IMID-Refractory Multiple Myeloma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unexpected toxicity (2 early deaths)
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201204086
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Bortezomib; carfilzomib; Dexamethasone; Cyclophosphamide; Thalidomide; Lenalidomide; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Filgrastim 5 ug/kg from Day -3 to Day 10 of a single cycle.
  Bortezomib will be given at the patient's current dose on Days 1, 4, 8, and 11 OR Carfilzomib will be given at the patient's current dose on Days 1, 2, 8, 9, 15, and 16 OR IMID will be given at the patient's current dose once daily on Days 1-21. Patients receiving an IMID (thalidomide, lenalidomide, or pomalidomide) as part of a bortezomib or carfilzomb regimen should continue the same scheduled as the current regimen.
  Dexamethasone should be continued at the same dose and schedule as the patient's current regimen.
  PO cyclophosphamide should be continued at the same dose and schedule as the patient's current regimen.
  Interventions: Drug: Filgrastim; Drug: Bortezomib; Drug: Carfilzomib; Drug: Dexamethasone; Drug: Cyclophosphamide; Drug: Thalidomide; Drug: Lenalidomide; Drug: Pomalidomide

INTERVENTIONS:
Drug: Filgrastim
  Other Names: G-CSF; Neupogen®; Granulocyte Colony-Stimulating Factor
Drug: Bortezomib
  Other Names: Velcade®
Drug: Carfilzomib
  Other Names: Kyprolis®
Drug: Dexamethasone
Drug: Cyclophosphamide
  Other Names: Cytoxan
Drug: Thalidomide
  Other Names: Thalomid
Drug: Lenalidomide
  Other Names: Revlimid
Drug: Pomalidomide
  Other Names: Pomalyst

SUMMARY:
Based on the pre-clinical data the investigators hypothesize that G-CSF treatment in patients with multiple myeloma will generate a 'hostile' bone marrow microenvironment for myeloma cells, depriving them of key support signals and rendering them more sensitive to chemotherapy. The investigators therefore propose to do an initial pilot study 1) to explore the safety of the combination of G-CSF and bortezomib-, carfilzomib-, or IMID-based treatment regimens in patients with bortezomib-, carfilzomib-, or IMID-refractory myeloma and 2) to generate correlative data for a subsequent larger study looking at the combination.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a confirmed diagnosis of multiple myeloma. The patient may be any stage of multiple myeloma. The patient may have received one or more lines of prior therapy (there is no limit to number of prior lines of therapy permissible).
* Patient must be ≥18 years of age
* Patient must be in active treatment with one of the following:

  * twice-weekly bortezomib (on Days 1, 4, 8, and 11 of a 21-day cycle) with or without dexamethasone
  * carfilzomib (on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle) with or without dexamethasone
  * an IMID with or without dexamethasone daily on Days 1 to 21.
  * Patients being treated with bortezomib or carfilzomb may also be receiving an IMID or PO cyclophosphamide with the regimen.
* Patient must have shown stable or progressive disease on the current bortezomib-, carfilzomib-, or IMID-containing regimen with a measurable monoclonal protein component in the serum (at least 0.5 g/dl on electrophoresis or 0.05 g/dl [50mg/dl] on serum-free-light-chain). Patients who had an initial response on the current bortezomib-, carfilzomib-, or IMID-containing regimen but now have stable (plateaued) disease are eligible.
* Patient must have an ECOG performance status of 0 - 2
* Patient must be receiving concurrent treatment with bisphosphonates, with one dose occurring within 30 days prior to first day (Day -3) of protocol treatment
* Patient must have acceptable hematologic parameters, defined as:

  * Absolute neutrophil count > 1000 cells/mm3
  * Platelets ≥ 50,000 cells/mm3
  * Hemoglobin ≥ 8 g/dl
* Patient must have adequate liver function, defined as:

  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x upper limit of normal
  * Total bilirubin < 2 x upper limit of normal
* Patient must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Patient must not be receiving any agents with known or suspected anti-myeloma activity (other than bortezomib, carfilzomib, dexamethasone, an IMID or PO cyclophosphamide, and bisphosphonates with the current regimen)
* Patient must not be actively using myeloid growth factors
* Patient must not have had any prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, or other cancer from which the subject has been disease-free for at least 2 years
* Patient must not have any uncontrolled medical problems such as diabetes mellitus, coronary artery disease, hypertension, unstable angina, arrhythmias, pulmonary disease, and symptomatic heart failure
* Patient must not have neuropathy ≥ grade 3 or painful neuropathy ≥ grade 2 (NCI CTCAE v 4.0)
* Patient must not have any known active infections requiring IV antibiotic, antiviral, or antifungal therapy
* Patient must not be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety of the combination of G-CSF and bortezomib-, carfilzomib-, or IMID-based treatment regimens in patients with refractory multiple myeloma. | Up to 30 days after last treatment
  Number and grade of adverse events based on NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Effects of G-CSF on bone marrow and bone marrow cytokine and chemokine levels. Including: Quantification of marrow osteoblasts and CAR cells, measurement of SDF-1 (CXCL12), IL-6, BAFF, assessment of myeloma cell proliferation and survival in bone marrow | 14 days after last drug treatment
Response rate as defined by the International Myeloma Working Group (IMWG) criteria | 14 days after last drug treatment
Overall survival duration of patients treated on study | 1 year
  Defined as the date of first dose of study drug to the date of death from any cause.
Progression-free survival of patients treated on study | 1 year
  Defined as the interval from the date of first treatment to date of first documentation of disease progression.
Duration of response of patients treated on study | 1 year
  Defined as the interval from the date of first documentation of response to the first documentation of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu